CLINICAL TRIAL: NCT02826005
Title: Examination the Ability to Early Diagnose HCC
Brief Title: Examination the Ability to Early Diagnose HCC by Combining Three Biomarkers Technology Developed by WAKO, And Their Relevance to Cirrhotic of Patients With Various Backgrounds and the Israeli Population.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ilex Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: WAKOHCC2016
Record Dates: First submitted 2016-07-04; First posted 2016-07-07 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Fibrosis
MeSH Terms: conditions — Fibrosis

ARMS (2):
- cirrhotic patients (Experimental): if positive for 3 bio-markers- will be followed by MRI for HCC diagnosis
  Interventions: Device: MRI
- non cirrhotic patients (No Intervention): control group - 3 bio-markers will be measured only

INTERVENTIONS:
Device: MRI
  Arms: cirrhotic patients

SUMMARY:
Examination the ability to early diagnose HCC by combining three biomarkers technology developed by WAKO, And their relevance to cirrhotic of patients with various backgrounds and the Israeli population.

This blood test will serve as an additional diagnostic tool tools currently in use (Ultrasound and AFP levels) to cirrhotic patients with high risk to develop hepatocellular carcinoma.

Another group that will be examined for all three biomarkers will be patients which already diagnosed with hepatocellular carcinoma, and have normal AFP level in order to examine the correlation between the presence of tumor, the number of them and the tumor size and the three biomarkers concentration in their blood

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic liver disease or cirrhotic or with diagnoses HCC with HCV, HBV, NAFLD, Alcohol background

Exclusion Criteria:

* patients with chronic liver disease or cirrhotic or with diagnoses HCC with autoimmune background or other background than HCV, HBV, NAFLD and Alcohol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of HCC in cirrhotic patients with positive values of the bio-markers by MRI | within 3 years from the bio-markers examination